CLINICAL TRIAL: NCT02188251
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Study Investigating the Effects of Activamp on Body Weight, Fat Loss, and Metabolic Markers in Healthy Overweight Participants
Brief Title: A Study Investigating the Effects of Activamp on Body Weight, Fat Loss, and Metabolic Markers in Healthy Overweight Participants
Acronym: 14AWHG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Gencor Pacific Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 14AWHG
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Body Weight
Keywords: Activamp; Gynostemma pentaphyllum; Body weight; Fat Loss; Metabolic markers; Overweight participants; DXA; AMPK
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Activamp (Experimental): Capsules containing 225mg of Activamp (Gynostemma pentaphyllum extract), 1 capsule taken twice daily for 12 weeks
  Interventions: Dietary Supplement: Activamp
- Placebo (Placebo Comparator): 1 capsule taken twice daily for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Activamp
  Arms: Activamp
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of Activamp, a product containing gynostemma pentaphyllum extract, on body weight, fat loss and metabolic markers in healthy overweight adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female 21-55 years of age
* BMI of 25.0 kg/m2 to 29.9 kg/m2 (± 1.0kg/m2)
* Must have negative urine pregnancy test at screening
* Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result.
* Subject agrees to maintain their normal level of physical activity throughout the study
* Weight has been stable for the last 3 months
* Subject agrees to comply with study procedures
* Healthy as determined by laboratory results, medical history and physical exam
* Subject agrees not to participate in structured activity including resistance training and aerobic exercise more than 3 times per week
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Subject who have experienced a greater than 10% variation in body weight in the past 3 months
* History of, or current diagnosis of any major diseases of the cardiovascular, hepatic, renal, gastrointestinal, pulmonary or endocrine systems
* History of surgery for weight loss (including gastric bypass or lapband)
* History of conditions that could interfere with the test product or impede its absorption such as gastrointestinal disease (Crohn's disease) or experienced surgery (caecum or enterocele surgery)
* Subjects diagnosed with Type II Diabetes
* Subjects with active cancer (excluding basal cell carcinoma)
* Subjects with active eating disorders
* Subjects who have undergone anti-psychotic drug therapy within the past 2 months
* Use of prescription or over the counter medications known to affect weight within 3 weeks of randomization or during the study
* Use of any supplements, programs, or meal replacement products, other than those provided, intended to alter body weight within two weeks of screening or during the course of the study
* Use of illicit drugs or history of drug or alcohol abuse within the past 6 months
* Currently having more than 2 standard alcoholic drinks per day
* Participation in a clinical research trial within 30 days prior to randomization
* Allergy or sensitivity to test article ingredients
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Abnormal lab test results or any other medical or psychological condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline to week 12

SECONDARY OUTCOMES:
Change in calculated BMI | baseline to week 12
Change in calculated percent body fat | Baseline to week 12
Change in calculated body fat mass | Baseline to week 12
Change in calculated lean body mass | Baseline to week 12
Change in total body fat percentage | Baseline to week 12
  As determined by DXA scan
Change in total fat mass | Baseline to week 12
  As determined by DXA scan
Change in total lean mass | Baseline to week 12
  As determined by DXA scan
Change in percent android fat | Baseline to week 12
  As determined by DXA scan
Change in percent gynoid fat | Baseline to week 12
  As determined by DXA scan
Change in percent trunk and legs fat | Baseline to week 12
  As determined by DXA scan
Change in percent abdominal fat | Baseline to week 12
  As determined by DXA scan
Change in anthropometric measurements | Baseline to 12 weeks
  Waist and Hip circumference
Change in blood AMPK activity | Baseline to week 12
Change in blood metabolic parameters | Baseline to 12 weeks
  lipid profile, Apo A1, Apo B, FFA, insulin and glucose, HOMA-IR, HbA1c, IGF, HsCrp, TNFalpha and glycerol
Change in blood safety parameters | Baseline to week 12
  CBC, electrolytes, markers of kidney and liver function
Changes in safety vital signs | Baseline to week 12
  Blood pressure, heart rate
Incidence of adverse events | Baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Dale Wilson, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada